CLINICAL TRIAL: NCT00787670
Title: Impact of Gastric Bypass Surgery on Risk of CVD in Type 2 Diabetes Mellitus
Brief Title: Impact of GBS on CVD in Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00006703; 5K23DK075907-02 (NIH)
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
Keywords: Obese; Type 2 Diabetes Mellitus; Gastric Bypass surgery; Risk of cardiovascular diseases
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gastric Bypass Surgery (Experimental): Gastric Bypass Surgery consists of a laparoscopic approach and includes the creation of an isolated 10-15-ml proximal gastric pouch, a retro-colic, retro-gastric Roux-en-Y gastrojejunostomy with linear stapler technique, a 100-cm Roux-limb, a 30-cm biliopancreatic limb, and a stapled end-side enteroenterostomy.
  Interventions: Procedure: gastric bypass surgery
- Diabetes Support and Education (Active Comparator): Diabetes Support and Eduction. Subjects attend three educational/social support sessions for 1 year after enrollment. The educational sessions offered for diabetes support and education including informational sessions on diet/nutrition and exercise. These sessions are informational only and do not teach behavioral self-regulation skills. Different nutrition and exercise topics are covered each session. Education
  Interventions: Other: Diabetes Support and Education
- Tissue Control Group (Active Comparator): Tissue control group includes subjects who are undergoing other non-gastric bypass abdominal surgery. A pea size piece of omentum and subcutaneous fat will be collected.
  Interventions: Other: Tissue Control Group

INTERVENTIONS:
Other: Diabetes Support and Education — The subjects will attend three educational/social support sessions for 1 year after enrollment. The educational sessions include informational sessions on diet/nutrition and exercise. These sessions are informational and do not teach behavioral self-regulation skills.
  Arms: Diabetes Support and Education
Procedure: gastric bypass surgery — gastric bypass surgery to induce weight loss in obese patients with type 2 diabetes
  Arms: Gastric Bypass Surgery
Other: Tissue Control Group — During the abdominal surgery we would like to take 5 ml blood from the IV line and small pea-sized samples of the fat tissue just under the skin and around the stomach area. These samples will be stored so that we can compare these tissue with other patients.
  Arms: Tissue Control Group

SUMMARY:
This research is a NIH single site study with the aims to (1) determine whether surgically induced weight loss decreases the risk of CVD in morbidly obese subjects with T2DM. (2) elucidate the mechanisms by which surgically induced weight loss reduces over time the risk of CVD in morbidly obsess subjects with T2DM.

Study'subjects will be enrolled from obese individuals with type 2 diabetes (T2DM). The study includes two groups, subjects undergoing gastric bypass surgery and a control group not undergoing weight loss surgery. A total of 60 subjects (30 in each group) will be recruited.

Basal, 6 and 12 months assessments will include: insulin sensitivity determination, cardiovascular function by echo doppler, and DEXA scan.

This study involves risk-level II procedures, however, the risks inherent to the gastric bypass surgery are not considered study-derived because subjects are enrolled from individuals that have already decided to have this surgery. We will determine protein expression profiles of inflammation-related adipokines in the subcutaneous and intra-abdominal adipose tissues of morbidly obese subjects with T2DM before and after surgically induced weight loss.

DETAILED DESCRIPTION:
Patients with type 2 diabetes mellitus (T2DM) are more likely to die from cardiovascular diseases (CVD) than people without diabetes. Furthermore, Patients with diabetes have not benefited from the advances in the management of CVD and/or its risk factors that have resulted in a decrease in mortality for CVD patients without diabetes. Short-term studies have demonstrated that weight loss in over weight or obese subjects with T2DM is associated with decreased insulin resistance, substantial improvements in glycemic and lipoprotein profile, and reduction in blood pressure. However, Long-term data substantiating that these improvements can be maintained are limited. Obesity, and susceptibility to weight gain, is a chronic condition. Continuous care is required to avoid weight regain especially after intensive weigh loss. Morbidly obese patients with body mass index (BMI) over 35 kg/m2 have significant difficulties maintaining weight loss adequate to resolve obesity-related medical conditions by changes in lifestyle or pharmacologic strategies. Currently, surgical treatment of morbid obesity, termed bariatric surgery, appears to be the only modality that results in significant and sustained weight loss along with reversal of diabetes and improvements in cholesterol biosynthesis, and lipoprotein metabolism in morbidly obese patients. Given these observations, we question if patients with T2DM who undergo gastric bypass surgery will significantly reduce levels of abnormalities in vascular structure and function that are central to the development of atherosclerosis. In specific aim 1, we will determine whether surgically induced weight loss decreases the risk of CVD in morbidly obese subjects with T2DM. . In specific aim 2, we will elucidate the mechanisms by which surgically induced weight loss reduces over time the risk of CVD in morbidly obsess subjects with T2DM. The proposed study is a prospective cohort clinic trial aimed to evaluate changes over time in cardiovascular structure and function of morbidly obese subjects with T2DM undergoing gastric bypass surgery compared to a matched control group who do not undergo gastric bypass surgery. The results of the proposed study will provide the foundation for a new clinic strategy aimed to prevent the development of CVD in obese patients with T2DM. Furthermore, it will serve as the baseline for future large scale longitudinal studies based on aggregate occurrence of severe cardiovascular events.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of T2DM diabetes mellitus with HbA1c ≤ 10.0%
* Current regular use of insulin
* Current regular use of oral hypoglycemic medication.
* Documented diabetes by current ADA criteria (98).
* Body mass index ≥ 35 kg/m2 in accord with the 1991 NIH obesity surgery consensus conference criteria and stable weight for the previous 3 months
* Age between 18-60 years old.
* Ability and willingness to provide informed consent.
* No expectation that subject will be moving out of the area of the clinical center during the next 12 months.

Exclusion criteria:

* Presence of CVD defined as: CAD, electrocardiographic criteria for past myocardial infarction(s), ischemic stroke, peripheral artery bypass surgery, percutaneous transluminal angioplasty, or amputation because of atherosclerotic disease
* Significant non-diabetic co-morbidity affecting life expectancy (e.g., malignancy)
* Significant other co-morbidities (e.g. psychiatric disorder) that results in ineligibility for gastric bypass surgery
* Pregnancy or planning pregnancy
* Severe dyslipidemia (triglycerides >600 mg/dl or cholesterol >350 mg/dl)
* Uncontrolled hypertension
* Smoking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2008-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To determine whether surgically induced weight loss decreases the risk of CVD in morbidly obese subjects with Type 2 Diabetes Mellitus (T2DM) | 0, 6, 12 months
  Patients with T2DM who undergo gastric bypass surgery will significantly reduce mean levels of risk factors for CVD compared with diabetic individuals with the same BMI who maintain their weight.

SECONDARY OUTCOMES:
To elucidate the mechanisms by which surgically induced weight loss reduces over time the risk of CVD in morbidly obese subjects with T2DM. | 0, 6, 12 months
  The reduction in CVD risk is mediated by changes in the expression and release of inflammatory-related adipokines by the adipose tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Torquati, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health system, Durham, North Carolina, United States

REFERENCES:
- [Derived] Khoo CM, Chen J, Pamuklar Z, Torquati A. Effects of Roux-en-Y gastric bypass or diabetes support and education on insulin sensitivity and insulin secretion in morbidly obese patients with type 2 diabetes. Ann Surg. 2014 Mar;259(3):494-501. doi: 10.1097/SLA.0b013e318294d19c. PMID 23732262